CLINICAL TRIAL: NCT01424579
Title: Effectiveness of Diacutaneous Fibrolysis for the Treatment of Subacromial Impingement Syndrome: a Randomised Controlled Trial
Brief Title: Diacutaneous Fibrolysis and Subacromial Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIC-P07/22
Record Dates: First submitted 2011-08-24; First posted 2011-08-29 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Actual Diacutaneous Fibrolysis (Experimental): The group received tree weeks of a daily protocolized treatment and additionally six sessions (two a week) of actual Diacutaneous Fibrolysis.
  Interventions: Other: Actual Diacutaneous Fibrolysis; Other: Protocolized physiotherapeutic Treatment
- Placebo Diacutaneous Fybrolisis (Placebo Comparator): This group received tree weeks of a daily protocolized treatment and additionally six sessions (two a week) of placebo Diacutaneous Fibrolysis.
  Interventions: Other: Placebo Diactuaneous Fibrolysis; Other: Protocolized physiotherapeutic Treatment
- No Diacutaneous Fibrolysis (Other): This group received only tree weeks of a daily protocolized treatment.
  Interventions: Other: Protocolized physiotherapeutic Treatment

INTERVENTIONS:
Other: Actual Diacutaneous Fibrolysis — Diacutaneous Fibrolysis is a non-invasive physiotherapeutic technique applied by means of a set of metallic hooks ending in a spatula with bevelled edges that allow a deeper and more precise application, which could not be achieved manually. Appropriate hook is applied following the intermuscular septum between the muscles with an anatomical or functional relationship with the painful structure, in a centripetal direction towards the pain location, in order to release adherences between musculoskeletal structures.
  Arms: Actual Diacutaneous Fibrolysis
Other: Placebo Diactuaneous Fibrolysis — Placebo Diacutaneous Fibrolysis was applied at a superficial level and, instead of fibrolysis, a pinch of skin was held with the thumb of the palpatory hand and the tip of the spatula, without any action taking place on the deep tissular levels.
  Arms: Placebo Diacutaneous Fybrolisis
Other: Protocolized physiotherapeutic Treatment — Tree weeks of daily therapeutic exercises, analgesic electrotherapy and cryotherapy.

SUMMARY:
Subacromial Impingement Syndrome (SIS) is the most common cause of shoulder pain with high lifetime prevalence (one in three) in general population. In occupational population is the most common upper extremity disorder. Symptoms include pain, a variable degree of mobility limitation and a more or less pronounced functional impairment. Conservative treatment is usually the first therapeutic option and some physiotherapeutic techniques have proved its efficacy but nevertheless treatment remains challenging.

According to the investigators clinical experience, Diacutaneous Fibrolysis has a beneficial effect on patients suffering from SIS, but no one published clinical trial has evaluated this manual technique previously. The investigators hypothesis is that adding Diacutaneous Fibrolysis to a protocolized physiotherapeutic treatment can provide better outcomes. The investigators objective was to assess the effect of Diacutaneous Fibrolysis on pain, mobility and functional status in patients suffering from SIS.

A double-blind (patient and evaluator) randomized clinical trial was carried out in two public centres of Primary Health Care of the Spanish National Health System. The study protocol was approved by the Clinical Research Ethics Committee from the Jordi Gol Institute of Research in Primary Health Care and all the patients provided written consent.

A hundred and twenty patients with clinical diagnosis of SIS were included and randomly allocated to one of three groups. All groups received the same daily protocolized treatment based on therapeutic exercises, analgesic electrotherapy and cryotherapy during three weeks. Additionally, intervention group received six sessions (two a week) of actual Diacutaneous Fibrolysis; placebo group received six sessions (two a week) of placebo Diacutaneous Fibrolysis, while control group received only the protocolized treatment.

Pain intensity (VAS), active range of motion (flexion, abduction, extension, external and internal rotation) and functional status (Constant-Murley score) were measured in baseline, after the three weeks of treatment and three months after the end of treatment.

ELIGIBILITY:
Inclusion criteria:

* Over 18 years
* Diagnosed of Subacromial Impingement Syndrome
* Signed a written consent form.

Exclusion criteria:

* Damaged skin and/or cutaneous lesions in the shoulder area,
* A concomitant treatment with platelet antiaggregant agents
* Acute inflammatory conditions in the shoulder
* Previous shoulder surgery
* A pending litigation or court claim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in Pain intensity at 3 weeks and 3 months | Baseline -3 weeks - 3 months.
  Measure instrument: Visual Analogue Scale

SECONDARY OUTCOMES:
Changes from Baseline in Active Range of Motion at 3 weeks and 3 months | Baseline - 3 weeks - 3 months
  Flexion, extension, abduction and external rotation movement were measured with a universal double-armed goniometer, and results are expressed in degrees.
  For Internal rotation the distance between the position achieved by the tip of the thumb in the hand-behind-back test and the inferior tip of the spinous process of C7 was measured with a flexible metric tape and results are expressed in centimeters.
Changes from Baseline in Functional status at 3 weeks and 3 months | Baseline - 3 weeks - 3 months
  Measure instrument: Constant-Murley score

CONTACTS AND LOCATIONS:
Overall Officials: Martín Barra-López, PT, Principal Investigator — Institut Català de la Salut; Carlos López-de-Celis, DO, PT, Study Chair — Institut Català de la Salut; Gabriela Fernández-Jentsch, PT, Study Chair — Servicio Gallego de Salud
Locations (1):
- ICS Servei de Rehabilitació Sant Ildefons, Cornellà de Llobregat, Barcelona, Spain

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/23523255